CLINICAL TRIAL: NCT02119299
Title: A Prospective, Single Arm, Multicenter Study Evaluating the Safety and Weight Loss Efficacy of the SMART Device + DVD Weight Loss Education for Overweight and Obese Adults
Brief Title: Safety and Efficacy of the SMART Device for Overweight and Obese Adults
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scientific Intake Limited Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0007
Record Dates: First submitted 2014-03-21; First posted 2014-04-21 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SMART device (Experimental): Use of Sensor Monitored Alimentary Restriction Therapy (SMART) device
  Interventions: Device: SMART device

INTERVENTIONS:
Device: SMART device — Sensor Monitored Alimentary Restriction Therapy (SMART) device
  Other Names: Sensor Monitored Alimentary Restriction Therapy

SUMMARY:
The purpose of this study is to demonstrate that (1) we will observe at least 40% of the subjects in the Per Protocol population having a measured ≥5% weight loss at 16 weeks compared to week 0; and (2) the observed mean % Total Body Weight Loss at 16 weeks compared to Week 0 is ≥4% in the Per Protocol population.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing and able to sign an informed consent for the study and has signed the IRB approved Information and Consent form for this study.
* Subject is age 18 to 49 years inclusive.
* Subject has a BMI between 27 and 35 kg/m² inclusive. Subject reports weight has been stable (no increase or decrease of 3% or more) in the last 3 months.
* Subject reports that he/she has had a dental check-up within the last 12 months.
* Subject reports that he/she is under the care of a dentist or orthodontist that the HCP may contact and provides name and location of the dental professional.
* Subject able to participate fully in and for the full duration of the study.
* Subject agrees to sign a behavioral contract describing that they understand the mechanism by which the device reduces food intake, that they will use the device during all meals and eating episodes (including snacks and while consuming sugar-sweetened liquids), that they will properly care for the device and that they will attend all study visits.
* Subject is fully ambulatory.
* Subject has normal condition, anatomy and function of the oral cavity as self-reported and confirmed by the trained health care provider.
* If female, the subject is; a. not pregnant (or lactating), and b. using and will continue to use adequate contraception throughout participation in the study.
* Subject reports no functional problems when swallowing solids or liquids.
* Subject lives or works within 25 miles of the study site and has a reliable method of transportation.

Exclusion Criteria:

* Subject has participated in a weight loss program and/or in a formal weight loss program (commercial, licensed counselor-delivered or medically supervised) in the last three months preceding anticipated study entry.
* Subject reports history of, or current, clinically significant disease, including: cardiovascular, pulmonary, gastrointestinal, urological, dermatological, central or peripheral nervous system, or endocrine disease or condition (other than type 2 diabetes that does not require insulin or sulfonylurea).
* Subject has a history of bariatric surgery.
* In the opinion of the Investigator, subject has respiratory, dental, oral, or neurological disease or condition that might interfere with use or safety of the SMART device.
* Subject has compromised oral health (e.g., decay, infection, abscess, loose or cracked teeth, inflamed oral tissue, receding gums, and periodontal disease).
* Subject uses antipsychotic medication. If the subject is on a stable dose (3 months or more) of an antidepressant he/she can be enrolled in the study.
* Subject has type 1 or type 2 diabetes and is taking insulin or sulfonylurea.
* Subject has history of malignant disease, other than non-melanoma skin cancer diagnosed within the last five years and successfully treated.
* Subject has known allergy to any component of the SMART device.
* Subject is a current smoker or user of smokeless tobacco or nicotine gum.
* Subject has recent history of drug or alcohol abuse (in last 3 years).
* Subject is known to be HIV positive.
* Subject has been diagnosed with Sjogren's syndrome or chronic dry mouth
* Subject has any of the following conditions in the oral cavity that would preclude fitting and wearing the device: oral deformity, upper arch removable partial dentures, inadequate oral anatomy (e.g., 3 or more loose or missing teeth on the upper arch, molars or pre-molars either missing or worn down to within 4 mm above gum line, teeth with excessive convexity or undercuts that will make placement and removal of the device difficult, an oro-nasal fistula secondary to cleft palate, or a large torus palatinus), veneers, temporary crowns or recently placed osteointegrated dental implants, and any fixed orthodontic appliances (e.g., braces).
* Subject is unable to complete the mold-making process.
* Subject is currently involved in another clinical trial or intends to participate in one during the study period.
* Subjects are excluded if they report the following eating patterns that are less likely to be helped by the SMART device; diagnosis of night eating syndrome* (wakened by hunger and desire to eat at night); diagnosis of sleep eating* (unconscious eating while asleep); self-report of consumption of 32 or more ounces of sugar-sweetened beverages per day; self-report of extremely slow eating, such that family members and friends remark on the trait; self-report of a grazing eating pattern, defined as eating or snacking in more than 6 episodes per day.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H Longley, Study Director — Scientific Intake
Locations (4):
- United States (4):
  - Investigative Site, San Diego, California
  - Investigative Site, Waterbury, Connecticut
  - Investigative Site, Coral Gables, Florida
  - Investigative Site, Sugar Land, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, there were two screening visits prior to the run-in visit to assess subject eligibility and oral health. A total of 4 visits (2 screening visits, 1 run-in visit and 1 wash-out visit) were included prior to the baseline visit.
Period: Overall Study
Arm/Group | SMART Device
Started | 76
Completed | 67
Not Completed | 9
Not completed — Withdrawal by Subject | 7
Not completed — Lack of Efficacy | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | SMART Device
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 76
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving ≥5% Weight Loss at 16 Weeks Compared to Week 0
Time Frame: 16 weeks
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Device
Number analyzed (Participants) | 40
Participants | 12

2. Primary Outcome: Mean %Total Body Weight Loss (TBL) at 16 Weeks Compared to Week 0
Time Frame: 16 weeks
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: % TBL
Arm/Group | SMART Device
Number analyzed (Participants) | 40
% TBL | 2.93 (3.531)

3. Secondary Outcome: Mean Percentage Excess Weight Loss (EWL)
Time Frame: 16 weeks
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: percentage of excess weight loss
Arm/Group | SMART Device
Number analyzed (Participants) | 40
percentage of excess weight loss | 18.76 (24.51)

4. Secondary Outcome: Mean Absolute Weight Loss (kg)
Time Frame: 16 weeks
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Body weight (kg)
Arm/Group | SMART Device
Number analyzed (Participants) | 40
Body weight (kg) | 2.35 (2.99)

5. Secondary Outcome: Proportion of Subjects Achieving ≥4% Weight Loss
Time Frame: 16 weeks
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Device
Number analyzed (Participants) | 40
Participants | 16

6. Secondary Outcome: Proportion of Subjects Achieving ≥12% EWL
Time Frame: 16 weeks
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Device
Number analyzed (Participants) | 40
Participants | 24

7. Secondary Outcome: Percentage Total Body Loss and Treatment Compliance Correlation
Description: The measured relationship between SMART device usage and total weight loss.
Time Frame: 16 weeks
Population: Per Protocol Population
Measure: Number; unit: Pearson correlation
Arm/Group | SMART Device
Number analyzed (Participants) | 40
Pearson correlation | .025

8. Secondary Outcome: Device Compliance
Description: Device compliance is calculated as 100*(# Device Uses Since Visit 5)/(# eating episodes since Visit 5).
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: % of eating episodes with device use
Arm/Group | SMART Device
Number analyzed (Participants) | 40
% of eating episodes with device use | 69 (14.13)

ADVERSE EVENTS:
Arm/Group | SMART Device
Serious Adverse Events (participants affected / at risk) | 1/76
Other Adverse Events (participants affected / at risk) | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SMART Device (N=76)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Subject discontinued due to becoming pregnant during study.

LIMITATIONS AND CAVEATS:
Lower percentage of TBL reported due to initial endpoint specifications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days